CLINICAL TRIAL: NCT03031665
Title: Sex, Hormones and GABA in Stress Induced Anhedonia in Depression
Brief Title: Sex, Hormones and Gamma-Aminobutyric Acid (GABA) in Stress Induced Anhedonia in Depression
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2016P000693
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: GABA; Depression; Stress; Androgens
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current MDD: Subjects experiencing a current episode of Major Depressive Disorder.
- Remitted MDD: Subjects who have a history of Major Depressive Disorder, but have not had a depressive episode for at least two months.
- Control Subjects: Subjects who have no history of clinical depression or other psychological disorder.

SUMMARY:
Using an innovative multi-modal imaging approach, this study investigates the role of the neurochemical gamma-aminobutyric acid (GABA), brain activity, as well as hormones in understanding sex differences in Major Depressive Disorder (MDD). Further, the investigators will link these markers to symptoms of depression.

DETAILED DESCRIPTION:
The goals of this research are to investigate: (1) functional and neurochemical features associated with depression irrespective of clinical state; (2) moderating effects of hormones on stress circuitry in MDD; and (3) sex differences in symptoms. To this end, the study is enrolling adults with current depression and remitted depression, along with a control group of psychiatrically health adults. Participants will have an magnetic resonance imaging (MRI) exam involving multiple imaging techniques (functional, structural, spectroscopic) while performing computer-based tests. Additional questionnaires and tests will be done outside the scanner to assess current symptoms and hormone levels. The integration of laboratory-based measures of reward and stress sensitivity, with state-of-the-art imaging techniques and hormonal assessments promises to provide novel insights in the sex-dependent manifestation and pathophysiology of MDD.

ELIGIBILITY:
Inclusion Criteria for all participants.

* Males and females aged 18 through 25
* Capable of providing written informed consent, and fluent in English
* Right-handed
* Absence of any psychotropic medications for at least 2 weeks
* Female subjects will be scheduled to participate during the follicular phase of their menstrual cycle

Inclusion Criteria for "Current MDD" group:

* Meets inclusion criteria for all subjects, plus:
* Meets diagnostic criteria for a current episode of Major Depressive Disorder (MDD), as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

Inclusion Criteria for "Remitted MDD" group:

* Meets inclusion criteria for all subjects, plus:
* History of MDD as defined by DSM-5, but in remission for the past two months
* Absence of anxiety disorder for the past two months

Exclusion Criteria for all participants:

* History of psychiatric illnesses, other than depression or anxiety disorders among the Current MDD and Remitted MDD groups.
* History of psychotic episodes, suicidal ideation, or of electroconvulsive therapy (ECT) treatment
* Use of hormone replacement therapy, or of anabolic steroids.
* Use of hormonal contraceptives is permitted for female subjects only if the subject has regular menses
* Failure to meet any MRI safety requirements
* Serious or unstable medical illness, or history of neurological disease or damage
* History of use of cocaine, stimulants, or dopaminergic drugs
* History of substance use disorder or alcohol use disorder (as these terms are defined by DSM-5); except depressed subjects may have a history of 'Mild' substance/alcohol use disorder only if it ended as least 12 months ago.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults (ages 18 to 25).
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level-dependent (BOLD) activation in response to stress | Baseline.
  Region-specific BOLD activation in response to stress in hypothalamus, amygdala, medial prefrontal cortex, orbitofrontal cortex, anterior cingulate cortex, and hippocampus

SECONDARY OUTCOMES:
Network-specific effective connectivity | Baseline
  Region-specific resting state connectivity of two networks (1) hypothalamus and amygdala, with medial prefrontal cortex and orbitofrontal cortex; and (2) hypothalamus and amygdala, with hippocampus
GABA concentration | Baseline
  Region-specific GABA concentration measured in rostral anterior cingulate cortex and dorsolateral prefrontal cortex

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No